CLINICAL TRIAL: NCT01203124
Title: A Single-blind, Randomized, Placebo Controlled, Parallel-group, Adaptive-design Study to Investigate the Impact of Dose and Dosing Frequency of AZD8848 Administered Intranasally for up to 7 Days, on the Biomarker
Brief Title: A Study to Investigate the Impact of Dose and Dosing Frequency of AZD8848 on the Response on Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D0540C00016; 2010-022574-14 (EudraCT Number)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers
Keywords: Intranasal; Biomarker; Healthy; Effect of different doses and dosing regimens of AZD8848 on biomarkers; Effect different doses and dosing frequency of AZD8848 on biomarkers
MeSH Terms: interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Placebo Comparator): Placebo given once daily on 7 days
  Interventions: Drug: Placebo
- 2 (Experimental): Active treatment at Day 1 and Day 7. Placebo on Day 2, 3, 4, 5 and 6
  Interventions: Drug: AZD8848; Drug: Placebo
- 3 (Experimental): Active treatment at Day 1, 4 and 7. Placebo on Day 2, 3, 5 and 6.
  Interventions: Drug: AZD8848; Drug: Placebo
- 4 (Experimental): Active treatment at Day 1, 3, 5 and 7. Placebo on Day 2, 4 and 6.
  Interventions: Drug: AZD8848; Drug: Placebo
- 5 (Experimental): Active treatment once daily on 7 days
  Interventions: Drug: AZD8848

INTERVENTIONS:
Drug: AZD8848 — The subjects are dosed with a range of intranasal doses of AZD8848 on 2, 3, 4 or 7 days of the 7 days treatment period. On the other days the subjects receive placebo.
  Arms: 2; 3; 4; 5
Drug: Placebo — Placebo
  Arms: 1; 2; 3; 4

SUMMARY:
The study will investigate how the dose of AZD8848 and the dosing frequency will affect the immunological/inflammatory response by measuring the production of biomarkers in blood and nasal lavage.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 55 years (inclusive). Women must be of non-childbearing potential or must have been stable on a highly effective contraceptive method for at least 3 months prior to Visit 1 and be willing to continue on the chosen contraceptive method, with additional use of a condom by male partners, until 3 months after last dose.
* Female subjects should have a negative pregnancy test at Visit 2 and date of last menstruation consistent of non-pregnancy
* Ability to metabolise AZD8848 (an in vitro screening assay will determine metabolic activity in a blood sample taken at Visit 1 using a pre-defined limit)

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings in physical examination
* Structural abnormalities of the nose or nasal disorder symptomatic enough to cause significant nasal obstruction
* Ongoing pregnancy or lactation
* Abnormal immune function

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2010-11; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
CXCL 10 (IP-10) and mRNA expression of IFNα regulated genes in blood and nasal lavage | Samples collected pre-dose and 1 day after first dose.
CXCL 10 (IP-10) and mRNA expression of IFNα regulated genes in blood and nasal lavage | Samples collected pre-dose and 7 days after first dose.
CXCL 10 (IP-10) and mRNA expression of IFNα regulated genes in blood and nasal lavage | Samples collected pre-dose and 8 days after first dose.
CXCL 10 (IP-10) and mRNA expression of IFNα regulated genes in blood and nasal lavage | Samples collected pre-dose and 10 days after first dose.
CXCL 10 (IP-10) and mRNA expression of IFNα regulated genes in blood and nasal lavage | Samples collected pre-dose and 12-14 days after first dose.

SECONDARY OUTCOMES:
To assess safety and tolerability of intranasal administration of AZD8848 at different doses and dosing regimens | During the 7 days dosing period and at four follow-up visits up to 11-13 months after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Leif T Eriksson, MD, PhD, Study Director — AstraZeneca; Wolfgang Kuhn, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1659&filename=D0540C00016_Study_Synopsis.pdf